CLINICAL TRIAL: NCT07346313
Title: The Effect of Reproductive Health And Sexual Rights Education Given to University Students With Escape Room Game on Sexual Health/Reproductive Health Knowledge Level And Perception of Gender Equality: A Randomized Controlled Study
Brief Title: The Effect of Escape Room Game on Reproductive Health Knowledge and Gender Equality Perception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karamanoğlu Mehmetbey University (Other)
Collaborators: Necmettin Erbakan University Scientific Research Projects Coordinator (Unknown); Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, GÜL BÜŞRA ALTUNAY DAVRAN, Lecturer, Karamanoğlu Mehmetbey University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: E-36321956-300-230705; 25DR9001 (Other Grant/Funding Number: Necmettin Erbakan Üniversitesi Bilimsel Araştırma Projeleri Koordinatörlüğü)
Record Dates: First submitted 2026-01-08; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Sexual Health; Reproductive Health; Gender Equality; Health Education
Keywords: Reproductive Health; Gender Equality; Gamification; Escape Room Game; Sexual Rights
MeSH Terms: conditions — Health Education | interventions — Gender Equity

STUDY DESIGN:
Intervention Model Description: This is a parallel-group randomized controlled study. Participants were randomly assigned into two separate groups: the intervention group and the control group. Both groups followed their respective protocols simultaneously over the same period, with the intervention group receiving an additional escape room educational module.
Masking Description: Since this is an educational intervention study, participants and investigators are aware of the group assignments. Therefore, masking is not applicable.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Both groups receive a standard theoretical education on reproductive health and family planning. Immediately following the educational session, the intervention group participates in the "Hidden Files in the Secret Laboratory" themed escape room game as an additional active learning module.
  Interventions: Behavioral: Escape Room Game on Reproductive Health and Gender Equality; Behavioral: Standard Theoretical Education
- Control Group (Active Comparator): This group receives the same standard theoretical education on reproductive health and family planning as the intervention group. To ensure educational equality and prepare all students equally for their final examinations, no additional game intervention is applied during the study period. However, to maintain ethical fairness, students in the control group are allowed to play the escape room game upon request after the post-test data collection is completed.
  Interventions: Behavioral: Standard Theoretical Education

INTERVENTIONS:
Behavioral: Escape Room Game on Reproductive Health and Gender Equality — A gamified educational intervention using an escape room format to teach reproductive health, sexual rights, and gender equality. Participants solve puzzles and complete tasks related to these topics within a set timeframe to improve their knowledge and perceptions.
  Arms: Intervention Group
Behavioral: Standard Theoretical Education — Standard theoretical education on reproductive health and family planning.

SUMMARY:
This study aims to evaluate the impact of an "escape room" educational game on university students' knowledge of sexual/reproductive health and their perceptions of gender equality. The research compares a group of students who received traditional theoretical education with a group that participated in an escape room game titled "Hidden Files in the Secret Laboratory" in addition to the same theoretical training. The primary goal is to determine if gamified learning enhances knowledge levels and shapes gender equality perceptions more effectively than standard education alone.

DETAILED DESCRIPTION:
This is a pretest-posttest, parallel-group, randomized controlled experimental study conducted at Karamanoğlu Mehmetbey University (2024-2025 Spring Semester).

The study population consists of 80 volunteer students enrolled in the Reproductive Health and Family Planning course, divided into two groups:

Intervention Group (n=40): Received standard theoretical education plus the "Hidden Files in the Secret Laboratory" themed escape room game.

Control Group (n=40): Received only the standard theoretical education.

Data collection was performed using a Descriptive Information Form, the Sexual Health and Reproductive Health Knowledge Scale, and the Gender Perception Scale. The study follows the CONSORT 2025 guidelines. Statistical analysis is performed using SPSS 26.0, including Chi-Square, ANOVA, and t-tests to compare pretest and posttest results between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older.
* Being proficient in the Turkish language.
* Enrolled in the "Reproductive Health and Family Planning" course for the first time.

Exclusion Criteria:

* Having any impairment that prevents effective communication (e.g., being a foreign national with insufficient Turkish reading/writing skills, or having hearing, speech, or cognitive disorders).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
Gender Perception Scale Score | Baseline (Pre-test) and 1 week after the intervention (Post-test).
  This scale evaluates the participants' perceptions of gender equality. It consists of multiple items rated on a Likert-type scale. Total scores are calculated, where higher scores reflect a more positive and egalitarian perception of gender roles.
Sexual Health and Reproductive Health Knowledge Scale Score | Baseline (Pre-test) and 1 week after the intervention (Post-test).
  This scale measures the participants' knowledge levels regarding sexual and reproductive health. The score is calculated based on correct answers to specific questions. Higher scores indicate a higher level of knowledge.

CONTACTS AND LOCATIONS:
Locations (1):
- Karamanoglu Mehmetbey Universty, Karaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared with other researchers to ensure the confidentiality and privacy of the student participants, as per the ethical approval and informed consent obtained for this study.